CLINICAL TRIAL: NCT02045953
Title: A Randomised, Open-Label, Four Period, Crossover Study to Assess the Systemic Exposure of Fluticasone Propionate From FLIXOTIDE™ 250 HFA pMDI and of Fluticasone Propionate and Salmeterol From SERETIDE™ 250/25 HFA pMDI When Given With the VENTOLIN Mini-Spacer Compared to the Aerochamber Plus Spacer in Healthy Subjects
Brief Title: A Study to Assess the Systemic Exposure of FLIXOTIDE™ (Fluticasone Propionate) and SERETIDE™ (Fluticasone Propionate and Salmeterol) Given With VENTOLIN™ Mini-Spacer Compared to the Aerochamber Plus Spacer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201092
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: Healthy Subjects; SERETIDE; Pharmocokinetics; FLIXOTIDE; VENTOLIN Mini-Spacer
MeSH Terms: conditions — Asthma | interventions — Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): Participant will receive study treatments in following sequence in four treatment periods (one treatment per period): ABCD, where A= FLIXOTIDE 250 Hydrofluoroalkane (HFA) with Aerochamber Plus spacer, B= FLIXOTIDE 250 HFA with VENTOLIN Mini-Spacer, C= SERETIDE 250/25 HFA with Aerochamber Plus spacer, D= SERETIDE 250/25 HFA with VENTOLIN Mini-Spacer
  Interventions: Device: VENTOLIN Mini-Spacer; Device: Aerochamber Plus spacer
- Sequence 2 (Experimental): Participant will receive study treatments in following sequence in four treatment periods (one treatment per period): BDAC, where A= FLIXOTIDE 250 HFA with Aerochamber Plus spacer, B= FLIXOTIDE 250 HFA with VENTOLIN Mini-Spacer, C= SERETIDE 250/25 HFA with Aerochamber Plus spacer, D= SERETIDE 250/25 HFA with VENTOLIN Mini-Spacer
  Interventions: Device: VENTOLIN Mini-Spacer; Device: Aerochamber Plus spacer
- Sequence 3 (Experimental): Participant will receive study treatments in following sequence in four treatment periods (one treatment per period): CADB, where A= FLIXOTIDE 250 HFA with Aerochamber Plus spacer, B= FLIXOTIDE 250 HFA with VENTOLIN Mini-Spacer, C= SERETIDE 250/25 HFA with Aerochamber Plus spacer, D= SERETIDE 250/25 HFA with VENTOLIN Mini-Spacer
  Interventions: Device: VENTOLIN Mini-Spacer; Device: Aerochamber Plus spacer
- Sequence 4 (Experimental): Participant will receive study treatments in following sequence in four treatment periods (one treatment per period): DCBA, where A= FLIXOTIDE 250 HFA with Aerochamber Plus spacer, B= FLIXOTIDE 250 HFA with VENTOLIN Mini-Spacer, C= SERETIDE 250/25 HFA with Aerochamber Plus spacer, D= SERETIDE 250/25 HFA with VENTOLIN Mini-Spacer
  Interventions: Device: VENTOLIN Mini-Spacer; Device: Aerochamber Plus spacer

INTERVENTIONS:
Device: VENTOLIN Mini-Spacer — VENTOLIN mini-spacer will be used to dispense the SERETIDE Evohaler and FLIXOTIDE Evohaler
Device: Aerochamber Plus spacer — Aerochamber Plus spacer will be used to dispense the SERETIDE Evohaler and FLIXOTIDE Evohaler

SUMMARY:
The VENTOLIN Mini-Spacer is being developed in order to support patients in the Emerging Markets and Asia Pacific regions who do not have access to affordable spacers. The aim of this exploratory study is to investigate whether the systemic exposure for fluticasone propionate (FP) and salmeterol observed with the VENTOLIN Mini-Spacer is comparable to the systemic exposure for FP and salmeterol observed with the Trudell Aerochamber Plus spacer for both FLIXOTIDE and SERETIDE Metered Dose Inhaler (MDI) products. There will be four study periods in the study and all participants will receive four study treatments during the study. The total duration of study including screening, treatment period, washout period, and follow-up period will be 58 days. Study is planned to enroll 20 healthy subjects.

VENTOLIN is a registered trademark of GlaxoSmithKline. FLIXOTIDE is a registered trademark of GlaxoSmithKline. SERETIDE is a registered trademark of GlaxoSmithKline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac testing. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and body mass index within the range 19 - 34 kg/meter^2 (inclusive).
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented hysterectomy, bilateral oophorectomy or bilateral salpingectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 21.7 international unit/Liter (L) and estradiol <110 picomoles/L is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.] Child-bearing potential with negative pregnancy test as determined by urine or serum human Chorionic Gonadotropin (hCG) test at screening or prior to dosing AND Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 2 days post-last dose.

OR has only same-sex partners, when this is her preferred and usual lifestyle.

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Agrees to provide written consent to have information entered into The Over-volunteering Prevention System "TOPS".
* Alanine aminotransferase, alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged QT duration corrected for heart rate by Fridericia's formula (QTcF) values of single electrocardiograms (ECGs) obtained over a brief recording period: QTcF <450 milliseconds (msec).

Exclusion Criteria

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Positive smoking breath test or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immuno virus antibody.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Loss of more than 400 mL of blood during the 3 months before the trial, e.g. as a blood donor.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs (except simple analgesics), including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids from 7 days prior to the first and subsequent doses of study medication and until collection of the last PK sample for that study period.
* The subject is unable to use the inhaler and spacer devices correctly after training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2014-03-13 (Actual); Study Completion 2014-03-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration versus time curve over 24 hours (AUC[0-24h]) for FP | Samples will be collected at: pre-dose, and 5 minutes (m), 10m, 30m, 45, 1 hour (h), 1.5h, 2h, 4h, 8h, 10h, 12 h, 16h and 24 h post dose in each period
  Blood samples will be collected for pharmacokinetic analysis of Fluticasone propionate at the time points indicated
Maximum observed plasma drug concentration (Cmax) for Salmeterol | Samples will be collected at: pre-dose, and 5 minutes (m), 10m, 30m, 45, 1 hour (h), 1.5h, 2h, 4h, 8h, 10h, 12 h, 16h and 24 h post dose in each period
  Blood samples will be collected for pharmacokinetic analysis of Salmeterol at the time points indicated

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) for FP | Samples will be collected at: pre-dose, and 5 minutes (m), 10m, 30m, 45, 1 hour (h), 1.5h, 2h, 4h, 8h, 10h, 12 h, 16h and 24 h post dose in each period
  Blood samples will be collected for pharmacokinetic analysis of Fluticasone at the time points indicated
Area under the plasma drug concentration versus time curve AUC (0-24h) for Salmeterol | Samples will be collected at: pre-dose, and 5 minutes (m), 10m, 30m, 45, 1 hour (h), 1.5h, 2h, 4h, 8h, 10h, 12 h, 16h and 24 h post dose in each period
  Blood samples will be collected for pharmacokinetic analysis of Salmeterol at the time points indicated
Time to maximum observed plasma drug concentration (tmax) for FP and Salmeterol | Samples will be collected at: pre-dose, and 5 minutes (m), 10m, 30m, 45, 1 hour (h), 1.5h, 2h, 4h, 8h, 10h, 12 h, 16h and 24 h post dose in each period
  Blood samples will be collected for pharmacokinetic analysis of Fluticasone propionate and Salmeterol at the time points indicated

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 201092 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201092?search=study&study_ids=201092#rs
- Available data/document: Individual Participant Data Set: 201092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201092 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register